CLINICAL TRIAL: NCT00001271
Title: A Phase I Study of Continuous Infusion Immunotoxin IgG-RFB4-SMPT-dgA in Refractory CD22 Positive B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 910176; 91-C-0176
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-06

CONDITIONS: B Cell Lymphoma
Keywords: Antigen Modulation; Pharmacokinetics; Ricin A Chain
MeSH Terms: conditions — Lymphoma, B-Cell

INTERVENTIONS:
Drug: IgG-RFB4-SMPT-dgA

SUMMARY:
Patients with CD22(+) B-cell lymphomas will be treated with escalating doses as a 192 hr infusion of immunotoxin in a Phase I study to determine dose limiting toxicity evidence of response.

DETAILED DESCRIPTION:
Patients with CD22(+) B-cell lymphomas will be treated with escalating doses as a 192 hr infusion of immunotoxin in a Phase I study to determine dose limiting toxicity evidence of response.

ELIGIBILITY:
Patients with a histologic diagnosis confirmed from a pretreatment biopsy at the Laboratory of Pathology, NCI of one of the following entities: Diffuse small Lymphocytic Lymphoma; Follicular, Small Cleaved cell Lymphoma; Follicular, Mixed Small Cleaved and Large Cell Lymphoma; Follicular Large Cell Lymphoma; Diffuse, Intermediately Differentiated Lymphocytic Lymphoma; Diffuse, Small Cleaved Cell Lymphoma; Diffuse, Mixed Small and Large Cell Lymphoma; Diffuse, Large Cell Lymphoma; Large Cell Immunoblastic Lymphoma; Small Noncleaved Cell Lymphoma.

Presence of CD22 antigen on at least 30 percent of tumor cells.

Presence of objectively measurable sites of disease. Bone marrow positivity and circulating tumor cells in the peripheral blood will be considered evaluable but not measurable disease.

No patients with purely B-cell Lymphosarcoma cell leukemia without nodal or soft tissue involvement.

No patients with B-cell chronic lymphocytic leukemia, or B-cell or pre-B-cell acute lymphocytic leukemia, and hairy cell leukemia.

Patients with objectively measurable disease outside a radiation port or disease which has clearly progressed within a radiation port.

HIV negative.

No CNS disease.

No pulmonary parenchymal disease.

Pleural effusions or ascites may be present.

Patients with progression of disease despite at least one standard combination chemotherapy regimen.

No chemotherapy for at least two weeks prior to entry.

Patients who do not desire or are not candidates for autologous or allogeneic bone marrow transplantation procedures.

Life expectancy of at least 3 months

Creatinine clearance greater than 60 cc per minute.

Total bilirubin less than 1.5 mg/dl.

SGPT less than 2 times the upper limit of normal.

Albumin greater than 75 percent of the lower limit of normal.

If prior treatment with doxorubicin, the radionuclide or echocardiogram ejection fraction shall be at least 35 percent.

Performance status 0-2.

Not in need of current radiation therapy to alleviate local problems.

No prior exposure to murine antibodies.

No need for current corticosteroid treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Start 1991-07; Study Completion 2001-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Vitetta ES, Fulton RJ, May RD, Till M, Uhr JW. Redesigning nature's poisons to create anti-tumor reagents. Science. 1987 Nov 20;238(4830):1098-104. doi: 10.1126/science.3317828.
- [Background] Thorpe PE, Detre SI, Foxwell BM, Brown AN, Skilleter DN, Wilson G, Forrester JA, Stirpe F. Modification of the carbohydrate in ricin with metaperiodate-cyanoborohydride mixtures. Effects on toxicity and in vivo distribution. Eur J Biochem. 1985 Feb 15;147(1):197-206. doi: 10.1111/j.1432-1033.1985.tb08737.x. PMID 2982609
- [Background] Shen GL, Li JL, Ghetie MA, Ghetie V, May RD, Till M, Brown AN, Relf M, Knowles P, Uhr JW, et al. Evaluation of four CD22 antibodies as ricin A chain-containing immunotoxins for the in vivo therapy of human B-cell leukemias and lymphomas. Int J Cancer. 1988 Nov 15;42(5):792-7. doi: 10.1002/ijc.2910420527. PMID 3263328